CLINICAL TRIAL: NCT00685373
Title: An Open-label, Long-term Safety and Efficacy Study of ACZ885 (Anti-interleukin-1β Monoclonal Antibody) Administered for at Least 6 Months in Patients With the Following Cryopyrin-associated Periodic Syndromes: Familial Cold Autoinflammatory Syndrome, Muckle-Wells Syndrome, or Neonatal Onset Multisystem Inflammatory Disease
Brief Title: Efficacy and Safety of ACZ885 in Patients With the Following Cryopyrin-associated Periodic Syndromes: Familial Cold Autoinflammatory Syndrome, Muckle-Wells Syndrome, or Neonatal Onset Multisystem Inflammatory Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885D2306
Record Dates: First submitted 2008-05-27; First posted 2008-05-28 (Estimated); Results first posted 2011-05-27 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Cryopyrin-Associated Periodic Syndromes; Familial Cold Autoinflammatory Syndrome; Muckle Wells Syndrome; Neonatal Onset Multisystem Inflammatory Disease
Keywords: Cryopyrin-associated periodic syndromes (CAPS):; Familial Cold Autoinflammatory Syndrome (FCAS),; Muckle-Wells Syndrome (MWS),; MWS with overlapping symptoms of Neonatal Onset Multisystem Inflammatory Disease (NOMID) or Neonatal Onset Multisystem Inflammatory Disease (NOMID),; children,; systemic autoinflammatory disease,; CIAS-1 gene,; NALP-3,; ACZ885,; human monoclonal anti-human interleukin-1beta (IL-1beta),; antibody,; autosomal dominant,; familial autoinflammatory syndrome
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Multiple Pterygium Syndrome, Autosomal Dominant | interventions — canakinumab

ARMS (1):
- Canakinumab (ACZ885) (Experimental): Subcutaneous injection every 8 weeks based on participant's body weight. Body weight >40 kilogram (kg): 150 milligrams (mg) per injection and body weight <= 40 kg: 2 mg/kg per injection. For participants who did not experience sufficient symptomatic relief, an up-titration to the dose and/or more frequent doses were permitted as per protocol.
  Interventions: Drug: Canakinumab (ACZ885)

INTERVENTIONS:
Drug: Canakinumab (ACZ885) — 6 mL glass vial containing 150 mg lyophilized Canakinumab reconstituted with water for a subcutaneous injection every 8 weeks. Dosage based on body weight.

SUMMARY:
This will provided long-term safety and efficacy data for ACZ885 (a fully human anti-interleukin-1β [anti-IL-1β] monoclonal antibody) given as an injection subcutaneously in patients who participated in the CACZ885A2102 (NCT00487708), CACZ885D2201 (NCT00685373) or CACZ885D2304(NCT00465985) studies or newly identified patients with the following cryopyrin-associated periodic syndromes: Familial Cold Autoinflammatory Syndrome, Muckle-Wells Syndrome or Neonatal Onset Multisystem Inflammatory Disease.

The duration of this study was 6 months with a maximum duration of 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients at least 3 years of age
2. Diagnosis of Familial Cold Autoinflammatory Syndrome, Muckle-Wells Syndrome or Neonatal Onset Multisystem Inflammatory Disease. Prior agreement between the Investigator and Novartis for study eligibility is required for patients who do not have a molecular diagnosis of NALP3 mutations available (either testing not performed, or testing performed but negative)upon study entry. For those patients who have not been molecularly tested for NALP3 mutations, molecular testing should be performed during the course of the study
3. For patients under anakinra therapy or any other investigational IL-1 blocking therapy, these treatments should be discontinued prior to the baseline visit.
4. Patients from the CACZ885A2102 study may enter this study. However, dosing at Visit 2 (Baseline Visit) can only occur if either 1) the patient is experiencing disease flare or 2) at least two months have elapsed from their last injection even in the absence of flare, whichever is earlier.
5. Patients who completed the CACZ885D2304 study may enter this study
6. Patients who completed the CACZ885D2201 study may enter this study
7. Patients who discontinued from the CACZ885A2102, CACZ885D2201 or CACZ885D2304 studies and for whom in the Investigator's judgment (with prior agreement from Novartis) continued treatment with ACZ885 in this study is considered appropriate.

Exclusion Criteria:

1. Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation with the exception of trials with anakinra, other investigational IL-1 blocking therapies, and/or ACZ885.
2. History of being immunocompromised, including a positive HIV at screening (ELISA and Western blot) test result.
3. A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test result is not allowed.
4. No live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose.
5. History of recurrent and/or evidence of active bacterial, fungal, or viral infections.
6. Positive tuberculin skin test reaction (PPD 5 tuberculin units or as according to local standard practice) (>= 5 mm induration) at 48 to 72 hours after administration at the screening visit or within 2 months prior to the screening visit. Patients who have a positive PPD skin test with a documentation of BCG vaccination, who are at low environmental risk for tuberculosis (TB) infection or reactivation, and have a negative chest X-ray can be included.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (6):
  - Little Rock Allergy and Asthma Clinic, Little Rock, Arkansas
  - UCSF School of Medicine, San Francisco, California
  - Allergy Center at Brookstone, Columbus, Georgia
  - Rush-Presbyterian St. Lukes Medical Center, Chicago, Illinois
  - Cleveland Clinic, Cleveland, Ohio
  - University of Wisconsin, Madison, Wisconsin
- Novartis Investigative Site, Laken, Belgium
- France (4):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpelier Cedex
  - Novartis Investigative site, Nantes
- Germany (6):
  - Novartis Investigative site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative site, Heidelberg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Marburg
  - Novartis Investigative site, Tübingen
- Novartis Investigative site, New Delhi, India
- Italy (5):
  - Novartis Investigative site, Genova
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Rome
  - Novartis Investigative Site, Trieste
- Spain (3):
  - Novartis Investigative Site, Madrid
  - Novartis Investigative site, Oviedo
  - Novartis Investigative Site, Vigo
- Novartis Investigative site, Istanbul, Turkey (Türkiye)
- Novartis Investigative site, London, United Kingdom

REFERENCES:
- [Derived] Kuemmerle-Deschner JB, Hachulla E, Cartwright R, Hawkins PN, Tran TA, Bader-Meunier B, Hoyer J, Gattorno M, Gul A, Smith J, Leslie KS, Jimenez S, Morell-Dubois S, Davis N, Patel N, Widmer A, Preiss R, Lachmann HJ. Two-year results from an open-label, multicentre, phase III study evaluating the safety and efficacy of canakinumab in patients with cryopyrin-associated periodic syndrome across different severity phenotypes. Ann Rheum Dis. 2011 Dec;70(12):2095-102. doi: 10.1136/ard.2011.152728. Epub 2011 Aug 21. PMID 21859692

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included participants previously enrolled in CACZ885A2102 (NCT00487708), CACZ885D2304 (NCT00465985) and ACZ885 naive patients.
Period: Overall Study
Arm/Group | Canakinumab (ACZ885)
Started | 166
Completed | 151
Not Completed | 15
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 5
Not completed — Lack of Efficacy | 3
Not completed — Condition no longer requires study drug | 1
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 166
Age, Customized [Number; unit: participants]
  >= 3 to < 18 years | 47
  >= 18 to < 41 years | 65
  >= 41 to < 75 years | 52
  >= 75 years | 2
Gender [Count of Participants; unit: Participants]
  Female | 97
  Male | 69
Disease Characteristics [Number; unit: participants]
  Muckle-Wells Syndrome | 103
  Familial Cold Autoinflammatory Syndrome | 30
  Neonatal Onset Multi-System Inflammatory Syndrome | 32
  Information Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events (AEs), Death, Serious Adverse Events (SAEs), Discontinuation of Study Drug Due to an AE, Infections and Infestations and Injection Site Reactions
Description: The number of participants with Adverse Events and Infections & Infestations are regardless of study drug relationship by primary system organ class preferred term equal and/or greater than 2% in any group. The number of participants with mild injection site reactions= mild reactions observed on at least one occasion but no moderate or severe reactions. The number of participants with moderate injection site reactions= moderate reactions observed on at least one occasion but no severe reactions.
Time Frame: 2 years depending on when the participant enters the study
Population: Safety Population defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 166
participants
  Adverse Event | 150
  Death | 0
  Serious Adverse Event | 18
  Discontinuation of study drug due to an AE | 4
  Infections and Infestations | 109
  Any Injection Site Reactions | 13
  Mild Injection Site Reactions | 11
  Moderate Injection Site Reactions | 2

2. Secondary Outcome: The Percentage of Participants Without Disease Relapse as Determined by the Physician's Global Assessment of Autoinflammatory Disease Activity, Assessment of Skin Disease and Inflammation Markers.
Description: Disease relapse following complete response is defined as inflammation markers: C-Reactive Protein (CRP) and/or Serum Amyloid A (SAA) result > 30 mg/L AND Physician's Global Assessment of Autoinflammatory Disease Activity > minimal or Physician's Global Assessment >= minimal AND Skin Disease Assessment > minimal.
  Physician's Global Assessment of Autoinflammatory Disease Activity and Skin Disease Assessment (urticarial skin rash) are completed by the investigator using a 5 point rating scale: absent, minimal, mild, moderate and severe.
Time Frame: Every 8 weeks during the course of the trial for at least 6 months with a maximum duration of 2 years
Population: Safety Population defined as all participants who had at least one dose of study drug and were included in the Relapse Assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 141
Percentage of participants | 90.1

3. Secondary Outcome: Immunogenicity of Canakinumab (ACZ885)
Description: The number of participants who tested positive for anti-ACZ885 antibodies using the Biacore Assay at the end of the study.
Time Frame: Every 8 weeks during the course of the trial for at least 6 months with a maximum duration of 2 years
Population: Safety Population defined as all participants who received at least one dose of study drug and were tested for anti-ACZ885 antibodies at the end of the study.
Measure: Number; unit: participants
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 156
participants | 0

4. Secondary Outcome: Pharmacokinetics
Description: Mean Clearance from serum in Liter per Day (CLD) in adult participants >=18, pediatric participants <18 with body weight >40 kg and pediatric participants <18 with body weight <=40 kg.
Time Frame: Every 8 weeks during the course of the trial for at least 6 months with a maximum duration of 2 years
Population: Safety population defined as all participants who received at least 1 dose of study drug. 3 participants were excluded because dosing information was not available at the time of analysis.
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | Canakinumab (ACZ885)
Number analyzed (Participants) | 163
L/day
  Adult Participants >= 18 years | 0.179 (0.084)
  Pediatric Participants <18 years and >40 kg | 0.180 (0.145)
  Pediatric Participants <18 years and <= 40 kg | 0.083 (0.033)

ADVERSE EVENTS:
Arm/Group | Canakinumab (ACZ885)
Serious Adverse Events (participants affected / at risk) | 18/166
Other Adverse Events (participants affected / at risk) | 124/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=166)
Muckle-Wells syndrome (Congenital, familial and genetic disorders) | 1
Radicular cyst (Gastrointestinal disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic tonsillitis (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Hepatitis C antibody positive (Investigations) | 1
Transaminases increased (Investigations) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Nerve root compression (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2
Depression (Psychiatric disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Miscarriage of partner (Social circumstances) | 1
Abortion induced (Surgical and medical procedures) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (ACZ885) (N=166)
Abdominal pain (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 16
Pyrexia (General disorders) | 18
Bronchitis (Infections and infestations) | 18
Gastroenteritis (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 48
Rhinitis (Infections and infestations) | 27
Upper respiratory tract infection (Infections and infestations) | 17
Fall (Injury, poisoning and procedural complications) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Headache (Nervous system disorders) | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.